CLINICAL TRIAL: NCT04132492
Title: AGNES - Aging Nephropathy Study, a Prospective Observational Cohort of Chronic Kidney Disease in Elderly Patients
Acronym: AGNES
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AGNES
Record Dates: First submitted 2019-10-07; First posted 2019-10-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; Elderly; Mortality; Renal Replacement Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no intervention — there is no intervention

SUMMARY:
With the aging population, a high prevalence of obesity, systemic arterial hypertension and diabetes mellitus, we are facing an increased incidence of elderly patients with chronic kidney disease (CKD) initiating renal replacement therapy. The correct diagnosis of CKD, the prognosis of the elderly patient with CKD, mainly comparing initiated dialysis vs. remaining in conservative treatment, the nutritional prognostic markers (sarcopenia), cardiovascular, mineral and bone metabolism, geriatric syndromes and sleep disorders are still debatable. Elderly patients are usually excluded from clinical trials and the scientific evidence is either scarce or based on retrospective data. Thus, the present study is a prospective cohort to evaluate the long-term evolution of patients ≥ 70 years with stage 4 or 5 CKD. The main outcomes are mortality and dialysis as a combined event. These endpoints will be correlated with independent parameters: Klotho, FGF23, nutrition and sleep quality. Confounders variables are cognition, depression, demographic, clinical and laboratory parameters, and daytime somnolence. Patients will be followed at the nephrology outpatient clinic of the Hospital das Clinicas, Universidade de Sao Paulo. The sample size was calculated to be 200 subjects. The summary methodology will include a broad geriatric assessment, cognition test, fragility, Charlson comorbidity scores, biochemical measurements of urea, creatinine, alkaline phosphatase, parathyroid hormone, calcium, phosphorus, vitamin D, vitamin B12, folic acid, thyroid hormones, hepatitis virus, serum albumin, albumin/creatinine ratio, protein/creatinine ratio, 24-h urinary protein, Epworth Sleepiness Scale, Pittsburgh questionnaire, segmental electric bioimpedance, and nutritional evaluation by 24h dietary interview.

DETAILED DESCRIPTION:
Main outcome: combined event mortality-dialysis

Independent variables: nutrition status, sleep quality, Klotho and FGF-23 Confounders: clinical and demographic variables, Charlson comorbidity index, Laboratory parameters, depression, functionality, cognition.

ELIGIBILITY:
* Clinical diagnosis of Chronic Kidney Disease stage 4 or 5
* Minimal age of 70 years
* Must be able to understand and sign the consent form

Exclusion Criteria:

* Patients who did not accept and sign the consent form
* Patients with cancer and life expectance lower than 6 months
* Moderate to advanced dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Outpatients with CKD that have been followed in the nephrology service - Nephrogeriatric ambulatory
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Combined events mortality-dialysis | through study completion, an average of 2 years
  dialysis or death

CONTACTS AND LOCATIONS:
Overall Officials: Rosilene Elias, MD, Ph.D., Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Hospital das Clinicas, São Paulo, São Paulo
  - Unersidade de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coelho VA, Santos GG, Avesani CM, Bezerra CIL, Silva LCA, Lauar JC, Lindholm B, Stenvinkel P, Jacob-Filho W, Noronha IL, Zatz R, Moyses RMA, Elias RM. Design and methodology of the Aging Nephropathy Study (AGNES): a prospective cohort study of elderly patients with chronic kidney disease. BMC Nephrol. 2020 Nov 7;21(1):461. doi: 10.1186/s12882-020-02116-w. PMID 33160321